CLINICAL TRIAL: NCT02519582
Title: Phase II Trial to Investigate the Safety and Efficacy of Orally Applied Niclosamide in Patients With Metachronous or Synchronous Metastases of a Colorectal Cancer Progressing After Therapy
Brief Title: Drug Trial to Investigate the Safety and Efficacy of Niclosamide Tablets in Patients With Metastases of a Colorectal Cancer Progressing After Therapy
Acronym: Nikolo
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Center for Molecular Medicine (Other)
Responsible Party: Principal Investigator, Susen Burock, MD, Charite University, Berlin, Germany
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCCC-mCRC-01
Record Dates: First submitted 2015-07-30; First posted 2015-08-11 (Estimated); Last update posted 2018-09-12 (Actual); Status verified 2018-09

CONDITIONS: Colorectal Cancer
Keywords: Colorectal Cancer; S100A4
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Niclosamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Niclosamid (Experimental): Patients receive 2 g niclosamide orally per day until progression or toxicity
  Interventions: Drug: Niclosamide

INTERVENTIONS:
Drug: Niclosamide — 2 g per day orally

SUMMARY:
Phase II trial evaluating the safety and efficacy of oral appliqued niclosamide in patients who are progressive with metachronous or synchronous metastases of colorectal cancer among the previous therapy (Nikolo). Monocentric open-label clinical trial of phase II. All patients received 2 g p.o. niclosamide daily until progression (according to RECIST) or unacceptable toxicity or discontinuation of study for other reasons.

DETAILED DESCRIPTION:
Effectiveness:

• effectiveness is measured by progression-free survival evaluated by RECIST (Response Evaluation Criteria In Solid tumor).

Overall survival For overall survival, the curves are estimated using the Kaplan-Meier method

ELIGIBILITY:
Inclusion Criteria:

* Patient with metachronous or synchronous metastases of a colorectal cancer progression under standard therapy
* no proven brain metastases
* no curative option
* no standard therapy available
* Age > 18 years
* At least one metastases measurable according to Response Evaluation Criteria In Solid Tumors V 1.1 in CT or MRI scan not older than 2 weeks before inclusion into the trial
* Lab values within the usual borders for these patient group e.g.
* Neutrophil ≥ 1.5x109/ •Platelets ≥ 100x109/L
* Leukocytes ≥ 1.0x109/L
* Hemoglobin ≥ 9.0 g/dL or 5.59 mmol/l
* Bilirubin ≤ 2 x Upper Limit of Normal (ULN) if not due to Gilbert's syndrome
* Aspartate Aminotransferase ≤ 2.5x Upper Limit of Normal in patients without liver metastases or ≤ 5.0x Upper Limit of Normal in patients with liver metastases
* Alanine aminotransferase ≤ 2.5x Upper Limit of Normal in patients without liver metastases < 5.0 x Upper Limit of Normal in patients with liver metastases
* adequate renal function (creatinin ≤ 1.5x Upper Limit of Normal)
* Eastern Cooperative Oncology Group 0 - 1
* EKG without clinical significant abnormalities
* No other malignant disease (except colorectal cancer) within the last 5 years before inclusion in the trial except adequately treated basal cell carcinoma of the skin or squamous cell carcinoma of the skin, in situ carcinoma of the cervix. Patients with a malignant disease in history have to be free of disease for 5 years.
* No clinical significant heart disease like e.g.
* Uncontrolled blood pressure
* Heart failure New York Heart Association grade > 2
* Cardiac infarction within the last 12 months
* No known uncontrolled concomitant disease despite treatment like e.g.
* Chronic obstructive pulmonary disease (COPD)
* Serious infections
* No known alcohol or drug abuses
* Absence of any psychological, familial, sociological or geographical condition, potentially hampering compliance with the study protocol and follow-up schedule
* Patients should use adequate birth control measures, during the study treatment period and for at least 3 months after the last study treatment.
* For women of childbearing potential (WOCBP):negative pregnancy test 72 hours before the application of the first dose if the study drug
* Patients who are breastfeeding must stop breastfeeding before the first dose of the study drug and not restart till 8 week after the last drug intake.
* Written informed consent before inclusion according to the International Conference on Harmonisation good clinical practice (ICH GCP) and national/local regulations

Exclusion Criteria:

* Life expectancy < 3 months
* Participation in another interventional study within the last 30 days
* Known hypersensitivity against a part of the study drug
* Pregnancy or breastfeeding
* HIV infection oder active hepatitis B/C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2015-08; Primary Completion 2019-12 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | At 4 months
  defined as the time from patient inclusion to the date of progression

SECONDARY OUTCOMES:
Overall survival | From date of randomization until the date of death, assessed up to 2 years
  defined as the time from patient inclusion to the date of death or date of last follow-up news (censured data)
Time to progression | From date of randomization until the date of first documented progression, assessed up to 2 years
  Progression according to RECIST
Disease control rate | From date of randomization, assessed up to 2 years
  remission + partial remission + stable disease
Number of Adverse Events > grade 2 toxicities according to NCI Common Toxicity Criteria for Adverse Effects v 4.03 | From date of randomization, assessed up to 1 months after end ot therapy
  number of adverse events > grade 2 toxicities according to NCI Common Toxicity Criteria for Adverse Effects v 4.03
Number of Serious Adverse Events | From date of randomization, assessed up to 1 months after end ot therapy
  number of serious adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Charité Universitätsmedizin Berlin; Charité Comprehensive Cancer Center, Berlin, Germany

REFERENCES:
- [Derived] Burock S, Daum S, Keilholz U, Neumann K, Walther W, Stein U. Phase II trial to investigate the safety and efficacy of orally applied niclosamide in patients with metachronous or sychronous metastases of a colorectal cancer progressing after therapy: the NIKOLO trial. BMC Cancer. 2018 Mar 15;18(1):297. doi: 10.1186/s12885-018-4197-9. PMID 29544454